CLINICAL TRIAL: NCT01081288
Title: Nationwide Cluster-randomised Trial of Extending the NHS Breast Screening Age Range in England
Brief Title: Extending the National Health Service (NHS) Breast Screening Age Range
Acronym: AgeX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Principal Investigator, DrToralGathani, Associate Professor and Consultant Surgeon, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10/H0710/9
Record Dates: First submitted 2010-03-03; First posted 2010-03-05 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer Mortality
Keywords: Breast cancer; Breast screening; Mammography; Routine screening programme
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Women aged 47-49 invited for breast screening (Active Comparator)
  Interventions: Other: Invitation for breast screening
- Women aged 71-73 invited for breast screening (Active Comparator)
  Interventions: Other: Invitation for breast screening

INTERVENTIONS:
Other: Invitation for breast screening — Invitation for breast screening to women in different age groups

SUMMARY:
Nationwide cluster-randomised trial of extending the NHS breast screening age range in England

DETAILED DESCRIPTION:
In 1988, the national Breast Screening Programme (BSP) began offering women aged 50-64 years triennial mammographic screening and full national coverage was achieved by the mid-1990s.

In 2003, the age range for triennial screening was extended from 50-64 to 50-70 years; proposals from committees in the Department of Health to randomise this age extension and thereby to obtain reliable information on both the risks and benefits of additional screening at ages 65-70 were not adopted.

Currently, 80 breast screening units cover all of England, each responsible for a defined area, and each year they invite about 2.8 million women aged 50-70, with 2.0 million accepting. The BSP sets standards for the screening units and monitors performance through its national quality assurance network.

In 2007, the Prime Minister announced plans for eventual extension to the range 47-73 years. This offered another opportunity to obtain reliable evidence about the effects of extending the age range of triennial screening. Hence, a trial of this age extension has begun, in which only half are offered extra screening, with the effects monitored through routinely collected NHS statistics.

Following a 2009-10 pilot study of the acceptability of cluster-randomisation of additional screening at ages 47-49 and 71-73 in 5 breast screening units, the AgeX trial extended recruitment to about five-sixths of the breast screening clinics in England, and this cluster-randomisation continues.

In 2011, the Government deferred the earliest possible date when screening would be extended to all women aged 47-73. Later, Public Health England (PHE, which is responsible for government screening programmes) stated that final decisions about extension of the age range would await the emergence of reliable evidence of its effects. The AgeX trial will eventually provide this.

In 2012, an independent panel set up by the Department of Health and the charity Cancer Research UK reported "The UK breast screening programmes [at ages 50-70] confer significant benefit and should continue…. The impact of breast screening outside the ages 50-69 years is very uncertain. The Panel supports the principle of the ongoing trial in the UK [AgeX] for randomising women under age 50 and above age 70 to be invited for breast screening".

Meanwhile, as female life expectancy is increasing, interest has grown in the possible advantages of continuing to screen women not just in their early 70s but throughout their 70s. The advantages and the disadvantages of continuing triennial screening after age 70 would be seen more clearly in a trial of 2 or 3 additional invitations (covering ages 71-76 or 71-79) than in a trial of just one.

In 2013 the All-Party Parliamentary Group on Breast Cancer in Older Women (APPG) said "Women are not routinely invited for breast screening past the age of 70 … the current 'age extension trial' [of screening past age 70] … should be extended past 73 to 76, and, if appropriate … further extended". In a separate report in 2015 the APPG reiterated this conclusion.

Although AgeX began as a trial of additional screening at ages 47-49 and at ages 71-73, it has therefore become a trial in which the older women allocated additional screening can, where resources are available, continue be invited triennially at ages 71-76 or at ages 71-79, thereby assessing the effects of continuing triennial screening for several years after age 70.

ELIGIBILITY:
Inclusion Criteria:

* Female, and
* Aged 47-49 years or 71-73 years, and
* In a Breast Screening Unit participating in the study. (All Breast Screening Units in England are expected to participate in the study with the exception of a few that use non-standard methods for creating screening batches).

Exclusion Criteria:

* Anyone not satisfying the inclusion criteria

Ages: 47 Years to 73 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000000 (Estimated)
Dates: Start 2009-06 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Breast cancer mortality | 17 years

SECONDARY OUTCOMES:
Breast cancer incidence, up to the same date that the primary outcome (breast cancer mortality) is reported | 17 years
Breast cancer treatments, including use of mastectomy, chemotherapy and radiotherapy, up to the same date that the primary outcome (breast cancer mortality) is reported | 17 years
All-cause mortality, up to the same date that the primary outcome (breast cancer mortality) is reported | 17 years

CONTACTS AND LOCATIONS:
Overall Officials: Toral Gathani, MD MBBS FRCS, Principal Investigator — University of Oxford
Locations (1):
- Cancer Epidemiology Unit, Richard Doll Building, University of Oxford, Roosevelt Drive, Oxford, United Kingdom

REFERENCES:
- See also: Breast Screening Programme Age Extension Trial — http://www.agex.uk/